CLINICAL TRIAL: NCT05368584
Title: Relationship Between Level of GPCR Autoantibodies and Cardiac Structure & Funtions Based on UCG and CMR
Status: Unknown | Type: Observational
Last Known Status: Active, not recruiting
Sponsor: Beijing Friendship Hospital (Other)
Responsible Party: Principal Investigator, Hongwei Li, MD, chief physician, Beijing Friendship Hospital
Other Study IDs: BFH-autoantibodies and STEMI
Record Dates: First submitted 2022-05-06; First posted 2022-05-10 (Actual); Last update posted 2022-05-10 (Actual); Status verified 2022-05

CONDITIONS: STEMI
Keywords: STEMI; GPCR; PCI
MeSH Terms: conditions — ST Elevation Myocardial Infarction

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
This study is a prospective cohort study，we want to observe the changes of different cardiovascular antibody levels in STEMI patients undergoing emergency PCI;and combined with different cardiovascular antibody levels and various indicators, evaluate the impact of ischemia-reperfusion injury and prognosis in STEMI patients after emergency PCI.

DETAILED DESCRIPTION:
This study mainly observed the changes of different cardiovascular antibody levels in STEMI patients undergoing emergency PCI by measuring autoantibodies; and the changes of autoantibodies in STEMI patients compared with coronary angiography-negative patients. At the same time, combined with different cardiovascular antibody levels and various indicators, the effect of ischemia-reperfusion injury and prognosis after emergency PCI in STEMI patients was evaluated. The correlation between autoantibody changes and imaging indicators in STEMI patients was evaluated by cardiac color Doppler ultrasound and CMR.

ELIGIBILITY:
Inclusion Criteria:

* STEMI patients meet the diagnostic criteria of "Guidelines for the Diagnosis and Treatment of Acute ST-segment Elevation Myocardial Infarction (2015)"; ②STMEI patients undergoing emergency PCI should undergo emergency PCI within 12 hours of onset at Beijing Friendship Hospital affiliated to Capital Medical University; ③ The selected patients were able to complete the MRI and STE examinations; ④ They agreed to be enrolled in the trial and signed the informed consent.

Exclusion Criteria:

* Past myocardial infarction or revascularization (PCI or CABG); ②Congestive heart failure LVEF<40%; ③Atrial fibrillation; ④Renal insufficiency (GFR<30 ml/min); disease; ⑥ rheumatic immune system disease; ⑦ malignant tumor; ⑧ claustrophobia; ⑨ contraindication to CMR;

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: ① Patients with acute ST-segment elevation myocardial infarction (STEMI) who underwent emergency PCI in Beijing Friendship Hospital (Xicheng District) affiliated to Capital Medical University. ②In the Beijing Friendship Hospital (Xicheng District) affiliated to Capital Medical University, coronary angiography showed negative coronary angiography in patients with non-coronary heart disease.
Sampling Method: Non-Probability Sample
Enrollment: 1 (Estimated)
Dates: Start 2022-05-07 (Actual); Primary Completion 2022-12 (Estimated); Study Completion 2022-12 (Estimated)

PRIMARY OUTCOMES:
β1-AA, β2-AA, α1-AA, M2-AA and AT1-AA OD values | Admission Baseline
  About 10ml of venous blood was collected on the second day of admission, serum was separated, and the OD values of β1-AA, β2-AA, α1-AA, M2-AA and AT1-AA were detected by ELISA.

CONTACTS AND LOCATIONS:
Locations (1):
- Beijing Friendship Hospital, Beijing, China